CLINICAL TRIAL: NCT02610738
Title: Junior KICk-OFF. Development and Pilot Evaluation of Structured Self-management Education Packages for Children 11 Years of Age and Under With Type 1 Diabetes, Their Parents and Carers.
Brief Title: Junior KICkOFF: Diabetes Education for Children Under 11 Years
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Children's NHS Foundation Trust (Other)
Collaborators: University of Sheffield (Other); University of Leeds (Other); University Hospitals of Derby and Burton NHS Foundation Trust (Other); Sheffield Hallam University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: SCH/14/036
Record Dates: First submitted 2015-04-30; First posted 2015-11-20 (Estimated); Last update posted 2020-01-03 (Actual); Status verified 2019-12

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Junior KICk-OFF education programme (Experimental): Participants will attend an age appropriate self management programme (Junior KICk-OFF) designed to improve their knowledge and understanding of type 1 diabetes
  Interventions: Behavioral: Junior KICk-OFF education programme

INTERVENTIONS:
Behavioral: Junior KICk-OFF education programme — The Junior KICk-OFF course is an age appropriate eduction course which aims to improve the understanding and knowledge of children with type 1 diabetes. It has been designed with school teachers and educationalists to meet the learning needs of children aged 4-11yrs
  Other Names: Educational package

SUMMARY:
The aim of this study is to develop educational packages for children of primary school age with type 1 diabetes and their parents, and to undertake a small scale feasibility study to allow evaluation of the curriculum. Paediatric diabetes teams in the United Kingdom currently deliver education using largely unevaluated teaching materials. By working with the education profession the investigators aim to develop packages which are based on recognised educational theory and practice. The investigators hope that use of these will result in better blood glucose control, reducing the risk of longterm diabetes complications such as eye and kidney disease.

DETAILED DESCRIPTION:
The aim of the study is to

1. To produce an educational curriculum and teaching material for three groups

   * Key stage one (KS1)(4-7 yrs)
   * Key stage two (KS2) (8-11 yrs)
   * Parents
2. To undertake pilot evaluation to establish

   * the feasibility of running the different education sessions, addressing access and other practical issues
   * the educational value of the packages produced with the aim of further refinement of the curriculum
   * the acceptability of the sessions to participants and parents
   * a process evaluation of the individual components of the packages
   * potential biomedical and psychological benefits, to provide data for a power calculation for a larger randomised controlled trial of the effectiveness of the educational package

The first phase of the project involves development of curriculum for the education of 4-11 yr old children with type 1 diabetes. Participants in key stage one will be taught a basic understanding of carbohydrate, exercise and insulin balance, hypoglycaemia and injections/pump basics and blood glucose testing. Older participants (Key stage two) will be taught similar topics but with increasing complexity appropriate to their age and understanding. The teaching will use approaches similar to those employed in schools and therefore the research team will work with primary school teachers and experts in education to ensure appropriate techniques and resources are employed. The focus of the education for parents will be to help them teach and encourage their children to develop their diabetes skills as they grow up.

The second phase of the project involves delivery of courses to each age group. The main focus of this will be to assess the acceptability of the curriculum. Feasibility in terms of practical arrangements, timing, use of resources etc will be examined. Feedback from an independent expert observer as well as from participants and educators will allow the curriculum to be assessed and adapted if necessary prior to larger scale study.

Some outcome measures are being examined. The investigators aim to assess whether older children's knowledge has changed pre and post course, whether diabetes self management within the family has altered and whether there is any impact on glycaemic control and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Child 4-11 years of age
* Attending primary school
* Type 1 diabetes> 1 yr duration

Exclusion Criteria:

* Non English speaking families
* Significant learning difficulties
* Co-morbidity likely to affect glycaemic control

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2 (Actual)
Dates: Start 2015-01; Primary Completion 2015-11-30 (Actual); Study Completion 2015-11-30 (Actual)

PRIMARY OUTCOMES:
Qualitative assessment of curriculum | post course- within 2 weeks
  Interviews with participants (parents and children) using semistructured interview schedule. Investigators will be seeking opinion about the usefulness of the course, whether any sections failed to meet their needs and whether they felt their self management behaviour around diabetes has been influenced
Educational evaluation through observation of junior KICk-OFF courses | during course delivery: three half days for keystage 1 children, three days for keystage 2 children
  An independent academic educationalist will observe course delivery and using a structured assessment sheet will assess fidelity with the curriculum, engagement of learners, assessment of learning needs and delivery of the curriculum.
Participant feedback on teaching | 3 days
  Written and verbal evaluation will be sought at end of each day of the course to assess immediate acceptability of the curriculum and identification of elements which are successful or otherwise

SECONDARY OUTCOMES:
Change in frequency of blood glucose testing | Change in number of tests for 4 weeks pre course and weekly for 3 months post course.
  Blood glucose meters are downloaded using Diasend software at all clinic visits. Analysis will record the total number of blood tests each week
Change in psychological outcomes: child participants in key stage two age group | baseline and 3 months post course
  Validated questionnaires - Pediatric Quality of Life Inventory (PedsQL-G and D)
Change in Knowledge assessment for key stage 2 children | pre course , 2 weeks and 3 months post course
  A quiz and practical assessment of knowledge has been developed for participants aged 8-10 yrs. By posing scenarios investigators will assess their knowledge and understanding of diabetes.
Change in HbA1c between baseline and 6 months | Measured within 2 weeks pre course and at 3 and 6 months post course
  HbA1c is a measure of glycaemic control which is recorded routinely in diabetes care. A sample will be collected in clinic or at baseline data collection.
change in blood glucose variability | 4 weeks pre course to 12 weeks post course
  Blood glucose meter download on DIASEND will be analysed for day to day variability
change in weekly mean blood glucose level | from 4 weeks pre course to 12 weeks post course
  Data will be extracted from the Diasend software of all blood glocuse readings on the particpant blood glucose meter
Change in Quality of life - of child as assessed by parent participants | baseline and 3 months
  parent participants will complete validated questionnaire :PedsQL generic and PedsQL diabetes questionnaire
Change in perceived stress - parent participants | baseline and 3 months
  Completion of validated perceived stress questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Kath Price, Principal Investigator — Investigator
Locations (1):
- Sheffield Children's NHS Foundation Trust, Sheffield, Sheffield (South Yorkshire District), United Kingdom